CLINICAL TRIAL: NCT05538611
Title: Evaluation of the Management Effect of "Special-general-practice-community-family" Chain Quality Control Model With General Practice Department as the Core in General Hospitals on Patients With Chronic Heart Failure
Brief Title: Effect Evaluation of Chain Quality Control Management on Patients With Heart Failure
Acronym: HF
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Liangying (Other)
Responsible Party: Sponsor-Investigator, Liangying, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2022 (023)
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure is a chronic disease that spans the home as well as the outpatient and hospital Settings and requires multidisciplinary, continuous disease management. Heart failure management emphasizes seamless connection from admission to return to the family, so as to improve the efficiency of resource use. Early preventive intervention, timely and reasonable drug treatment, integration of effective medical resources, and establishment of A sound and effective management model should be carried out for the population with high risk factors of heart failure (heart function stage A), so as to delay the occurrence and development of heart failure and further avoid the occurrence of malignant cardiovascular events. Therefore, this project aims to establish a "special-general-community-family" chain quality control model with the "general practice department" as the core for patients with chronic heart failure in general hospitals, so as to provide them with a full life cycle, multidimensional, concise and efficient quality control management.At present, the situation of heart failure prevention and treatment in China is grim and the challenge is huge. Heart failure complicated illness, drug dosage adjustment characteristics of professionalism, its emphasis on guide oriented treatment, and should pay attention to individual, need of specialized subject doctor, general practitioners, community doctors and family personal collaborative to maximize the optimal management of patients with chronic heart failure, follow the classification diagnosis and treatment, two-way referral is helpful to improve the long-term prognosis of patients with. At present, HF management has received increasing attention, how to choose a more reasonable, effective and economic management mode is still a problem of disagreement.

DETAILED DESCRIPTION:
At present, there is no unified and publicly recognized management model at home and abroad, and most studies only involve the use of one or a few measures, while the organic combined application of various measures is rarely reported. To enable patients to have a better quality of life and life, and to establish a standardized and suitable quality control management mode for heart failure is one of the hot topics in the cardiovascular field.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with BNP > 100ng/ml in laboratory examination or LVEF < 50% in ultrasound ECG; 2. Meeting the CHF diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Heart Failure 2018; 3. Patients with cardiac function stage A-C: stage A, patients with high risk factors for heart failure (hypertension, coronary heart disease, diabetes and obesity, metabolic syndrome, history of cardiotoxic drugs, history of alcoholism, history of rheumatic fever, family history of cardiomyopathy, etc.); In stage B, cardiac structural changes (left ventricular hypertrophy, asymptomatic valvular heart disease, previous myocardial infarction) were present; In stage C, the patient has structural changes in the heart and has symptoms and/or signs of heart failure (dyspnea, fluid retention, edema of both lower limbs, etc.) in the past or present; 4. Patients with NYHA (New York Cardiology Society) cardiac function grade I to IV; 5. Age > 18, both sexes; 6. No mental disorder, clear consciousness and normal communication; 7. Non-pregnant and lactating women;

Exclusion Criteria:

* 1. Severe valvular disease, pericardial disease, cardiomyopathy, congenital heart disease, acute myocardial infarction (within 4 weeks), cardiogenic shock, acute myocarditis, severe arrhythmia with hemodynamic changes; 2. Patients with pulmonary heart disease, pulmonary hypertension caused by acute and chronic pulmonary embolism, and stroke in the past six months; 3. Complicated with other serious acute and chronic diseases, such as liver and renal failure, respiratory failure, malignant tumor, diabetes with serious complications, hyperthyroidism, hypothyroidism and other serious endocrine diseases; Autoimmune diseases, etc.; 4. Pregnant or lactating women; 5. Patients with mental disorders or verbal communication or cognitive disorders; 6. patients with infectious diseases; 8. The residence area is not fixed, and it is difficult to complete the follow-up or loss of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It met the CHF diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Heart Failure 2018
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Trend of adverse cardiovascular events after chain management of heart failure in general practice | 2021.09-2023.09
  The incidence of adverse cardiovascular events in patients with heart failure after chain management in general practice has a significant downward trend

CONTACTS AND LOCATIONS:
Overall Officials: ying Liang, Principal Investigator — Belong to
Locations (1):
- Liangying, Jinan, Shandongsheng, China